CLINICAL TRIAL: NCT06474039
Title: The Efficacy of Fluticasone Furoate/Vilanterol/Umeclidinium Compared With Vilanterol/Umeclidinium in Reducing Air Trapping and Airway and Blood Cytokine Levels in COPD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor Dr., Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si344/2024
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment 1 (Experimental): Phase 1
  Interventions: Drug: Trelegy or Anoro
- Treatment 2 (Experimental): Phase 2
  Interventions: Drug: Trelegy or Anoro

INTERVENTIONS:
Drug: Trelegy or Anoro — Both drugs delivered via Ellipta device and blinded package appearance

SUMMARY:
This study aims to demonstrate the effects of triple therapy (ICS/LABA/LAMA) and dual bronchodilators (LAMA/LABA) on air trapping in the lungs' COPD patients and inflammatory mediators

ELIGIBILITY:
Inclusion Criteria:

* Patients who have met the criteria for COPD GOLD B defined by an exacerbation not more than 1 time in the last year prior to the study enrollment. These patients will be recruited in sequential sequence.
* Patients with COPD GOLD B are previously treated with either LAMA or LAMA/LABA or short-acting bronchodilators
* Patients who are able to provide informed consent.

Exclusion Criteria:

* - Concomitant with active and old pulmonary TB, lung cancer, bronchiectasis, lung fibrosis, destroyed lung, other malignancy, active heart diseases.
* Receiving long-term treatment with immunosuppressive drugs and systemic corticosteroids
* Being treated with triple therapy (ICS/LABA/LAMA)
* Being in terminally ill conditions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in lung volume | 4 weeks
  TLC, RV, RV/TLC, IOS

SECONDARY OUTCOMES:
Inflammatory cytokines | 4 weeks
  FENO, hs-CRP, sputum cell counts and differential counts

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong Maneechotesuwan, MD,PhD, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Respiratory Disease and TB, Siriraj Hospital, Bangkoknoi, BKK, Thailand

IPD SHARING:
Plan to Share IPD: No